CLINICAL TRIAL: NCT06085482
Title: A Single-Group, Open-Label, Single-Period, Phase 1 Study to Determine the Absolute Bioavailability of LY3502970 in Healthy Participants
Brief Title: A Phase I Study of LY3502970 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 18596; J2A-MC-GZGO (Other: Eli Lilly and Company)
Record Dates: First submitted 2023-10-10; First posted 2023-10-17 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Healthy
MeSH Terms: interventions — orforglipron

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- LY3502970 + [14C]-LY3502970 (Experimental): Single dose of LY3502970 administered orally followed by single dose of [¹⁴C]-LY3502970 administered intravenously (IV)
  Interventions: Drug: LY3502970; Drug: [14C]-LY3502970

INTERVENTIONS:
Drug: LY3502970 — Administered orally
Drug: [14C]-LY3502970 — Administered IV

SUMMARY:
The main purpose of this study is to evaluate how much of the study drug (LY3502970) and the radioactive substance 14C incorporated LY3502970 gets into the bloodstream, how its broken down, and how long it takes the body to get rid of it. The study will last up to approximately 9 weeks for each participant.

ELIGIBILITY:
Inclusion Criteria:

* Are overtly healthy as determined by medical evaluation
* Participants with body weight of 45 kilograms (kg) or more and body mass index within the range 18.5 to 35.0 kilograms per meter squared (kg/m²), inclusive
* Males who agree to use highly effective or effective methods of contraception and women not of childbearing potential may participate in this study

Exclusion Criteria:

* Participants who have known allergies to LY3502970, related compounds, or any components of the formulation
* Women who are lactating and women of child bearing potential (WOCBP) are excluded from the study
* Participants who regularly use known drugs of abuse or show positive findings on drug screen

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2023-10-19 (Actual); Primary Completion 2024-01-05 (Actual); Study Completion 2024-01-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Absolute bioavailability of LY3502970 | Predose up to 16 days postdose
  PK: Absolute bioavailability of LY3502970

SECONDARY OUTCOMES:
PK: Area Under the Curve Concentration Versus Time Curve From zero to Infinity (AUC [0-∞]) of Total Radioactivity | Predose up to 16 days postdose
  PK: AUC [0-∞] of Total Radioactivity
PK: AUC [0-∞] of [14C]-LY3502970 | Predose up to 16 days postdose
  PK: AUC [0-∞] of [14C]-LY3502970
PK: AUC [0-∞] of LY3502970 | Predose up to 16 days postdose
  PK: AUC [0-∞] of LY3502970
PK: Maximum Concentration (Cmax) of Total Radioactivity | Predose up to 16 days postdose
  PK: Cmax of Total Radioactivity
PK: Cmax of [14C]-LY3502970 | Predose up to 16 days postdose
  PK: Cmax of [14C]-LY3502970
PK: Cmax of LY3502970 | Predose up to 16 days postdose
  PK: Cmax of LY3502970

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No